CLINICAL TRIAL: NCT06448598
Title: Exercise as an Adjunctive Therapy for Patients on Maintenance Hemodiafiltration: A 6- Month Analysis
Brief Title: Exercise as an Adjunctive Therapy for Patients on Maintenance Hemodiafiltration
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Lyon College (Other)
Responsible Party: Principal Investigator, Mayron Faria de Oliveira, Principal Investigator, Federal University of São Paulo
Other Study IDs: 60256122.0.0000.5505
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Kidney Diseases
Keywords: hemodiafiltration; dialysis; exercise
MeSH Terms: conditions — Kidney Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise: he exercise group consisted of patients who participated in the exercise program, which involved twice-weekly sessions of aerobic exercises performed at 70% of maximum heart rate from a step test, as well as resistance exercises at 60% of one-repetition maximum strength. Within the exercise group, participants self-selected into either the intradialytic subgroup, where exercise was performed during their hemodiafiltration (HDF) sessions, or the interdialytic subgroup, where exercise took place on non-dialysis days.
  Interventions: Other: Exercise
- Control: The control group did not undergo any exercise intervention or physical evaluations with a physical therapist. Data collected from the control group pertained solely to dialysis adequacy measures such as Kt/V and urea reduction ratio (URR). This allowed for comparisons between the exercise and non-exercise groups in terms of dialysis efficiency.

INTERVENTIONS:
Other: Exercise — The exercise protocol involved twice-weekly sessions, with aerobic exercises performed at 70% of the maximum heart rate achieved during the step test, and resistance exercises at 60% of 1RM. Participants self-selected their exercise timing, either intradialytic (during HDF sessions) or interdialytic (on non-dialysis days). For the intradialytic group, exercise was seamlessly integrated into the HDF session, excluding the initial and final two hours of dialysis.
  Groups: Exercise

SUMMARY:
Patients with chronic kidney disease suffer from uremic toxin accumulation. Treatments with hemodiafiltration demonstrate the highest capacity for removing solutes, as well as improving mortality. While exercise has been proven as an adjunct therapy in patients on maintenance hemodialysis, little is known about the exercise influence in maintenance hemodiafiltration programs.

Methods: A retrospective observational study of chronic kidney disease patients at Fenix Nephrology group from 2021 until 2023. Patients were assessed at the start of the exercise program and after six months of rehabilitation. Physical tests included a step-test for endurance, handgrip and one-repetition maximum for muscle strength. The Kidney Disease Quality of Life Short Form evaluated patient-reported outcomes. Kt/V urea and urea reduction ratio were surrogates for hemodiafiltration adequacy. Patients carried out twice weekly aerobic exercises at 70% of the maximum heart rate during the step test, and resistance exercises at 60% of one-repetition maximum.

DETAILED DESCRIPTION:
The objectives of this study were twofold: first, to understand if hemodiafiltration (HDF) combined with exercise is a safe and effective treatment for patients with end-stage renal disease (ESRD/CKD 5D); and second, to explore the efficacy of exercise performed during dialysis sessions (intradialytic) versus between sessions (interdialytic).

The study employed a retrospective observational design, analyzing data from CKD 5D patients undergoing maintenance HDF at the Fenix Nephrology group between 2021 and 2023. Inclusion criteria stipulated that participants were aged 18 years or older, on HDF with optimized medication, and agreed to participate in the exercise program with at least 80% adherence. Assessments were conducted at baseline and after six months of rehabilitation, including a step-test for endurance, handgrip strength measurement, one-repetition maximum (1RM) test for muscle strength, and the Kidney Disease Quality of Life Short Form (KDQOL-SF) questionnaire. Kt/V and urea reduction ratio (URR) were used as surrogates for HDF adequacy.

The exercise protocol involved twice-weekly sessions, with aerobic exercises performed at 70% of the maximum heart rate achieved during the step test, and resistance exercises at 60% of 1RM. Participants self-selected their exercise timing, either intradialytic (during HDF sessions) or interdialytic (on non-dialysis days). For the intradialytic group, exercise was seamlessly integrated into the HDF session, excluding the initial and final two hours of dialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing maintenance hemodiafiltration (HDF)
* Optimized medication regimen
* Agreed to participate in the exercise program with at least 80% adherence

Exclusion Criteria:

* Patients who underwent kidney transplantation during the study period
* Patients with missing data
* Patients with exercise participation below 80% adherence
* Presence of comorbidities such as COPD, stroke, muscle weakness, or recent orthopedic surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients with end-stage renal disease (ESRD/CKD stage 5D) undergoing maintenance hemodiafiltration (HDF) at the Fenix Nephrology Group between 2021 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Exercise Intervention | 6 months
  Determine if hemodiafiltration (HDF) combined with exercise is a safe and effective treatment for patients with end-stage renal disease compared to controls.

SECONDARY OUTCOMES:
Inter- and intra-dialysis exercise intervention | 6 months
  Compare the efficacy of exercise performed during dialysis sessions (intradialytic) versus between sessions (interdialytic).

CONTACTS AND LOCATIONS:
Locations (1):
- Fenix Nefrologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
All data will be stored and only the manuscript results will be published.